CLINICAL TRIAL: NCT04928638
Title: Educational Intervention for Asthmatic and Allergic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Principal Investigator; PT; PhD, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DF0096UG
Record Dates: First submitted 2021-03-25; First posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Asthma; Allergy
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual educational intervention (Experimental): Educational intervention about the disease, the use of medication and the context of pandemic
  Interventions: Behavioral: Virtual educational intervention
- Written educational intervention (Experimental): Educacional intervention about the disease, the use of medication and the context of pandemic
  Interventions: Behavioral: Written educational intervention
- Control intervention (No Intervention): Control intervention

INTERVENTIONS:
Behavioral: Virtual educational intervention — Educational intervention about the disease, the use of medication and the context of pandemic
  Arms: Virtual educational intervention
Behavioral: Written educational intervention — Educational intervention about the disease, the use of medication and the context of pandemic
  Arms: Written educational intervention

SUMMARY:
Despite its importance, there are few studies that implement the use of new technologies in the approach to patients with asthma and allergy. Therefore, the objective of this study is to evaluate the effectiveness of a telematic educational intervention in patients with allergies and / or asthma

ELIGIBILITY:
Inclusion Criteria:

* Asthmatic and allergic patients

Exclusion Criteria:

* Cognitive impairment.
* Diagnose of autism spectrum disorder or severe intellectual disability
* Physical or functional impairment that limits the performance of evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-12 (Estimated); Primary Completion 2021-07-12 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Asthma knowledge questionnaire | Baseline
  Questionnaire to evaluate the knowledge about asthma. The questionnaire consists of 23 questions, some of them with several items. In total, there are 54 possible true / false / don't know answers. Each correct answer is given the value of one point and each incorrect or unknown answer a score of 0. Thus, the score that can be obtained in total is 0-54.
Asthma knowledge questionnaire | 1month
  Questionnaire to evaluate the knowledge about asthma. The questionnaire consists of 23 questions, some of them with several items. In total, there are 54 possible true / false / don't know answers. Each correct answer is given the value of one point and each incorrect or unknown answer a score of 0. Thus, the score that can be obtained in total is 0-54.
Allergic rhinitis knowledge questionnaire | Baseline
  Questionnaire to evaluate the knowledge about Allergic rhinitis. It includes 7 items. Patients have to answer true/false. Higher puntuation indicates better knowledge results.
Allergic rhinitis knowledge questionnaire | 1month
  Questionnaire to evaluate the knowledge about Allergic rhinitis. It includes 7 items. Patients have to answer true/false. Higher puntuation indicates better knowledge results.
Inhaler technique checklist | Baseline
  Checklist to evaluate the technique of inhaler. It contains several items that need to be checked. If the patient has a puntuation of 0-3 it is considered poor technique; If the patien has a puntuation of 4-5 it is considered the patient has a Moderate technique and if the patient has 6-7 points the technique is Good
Inhaler technique checklist | 1month
  Checklist to evaluate the technique of inhaler. It contains several items that need to be checked. If the patient has a puntuation of 0-3 it is considered poor technique; If the patien has a puntuation of 4-5 it is considered the patient has a Moderate technique and if the patient has 6-7 points the technique is Good
Knowledge of COVID | Baseline
  Questionnaire to evaluate the knowledge about COVID-19. It includes 12 items. Patients have to answer true/false. Higher puntuation indicates better knowledge results.
Knowledge of COVID | 1month
  Questionnaire to evaluate the knowledge about COVID-19. It includes 12 items. Patients have to answer true/false. Higher puntuation indicates better knowledge results.

SECONDARY OUTCOMES:
Asthma control questionnaire | Baseline
  A simple questionnaire to measure the adequacy of asthma control and change in asthma control which occurs either spontaneously or as a result of treatment. 7 items; 1 week recall (for items on symptoms and rescue inhaler use). 7-point scale (0=no impairment, 6= maximum impairment for symptoms and rescue use; and 7 categories for FEV1%). Minimally important difference: Change in score of 0.5
Asthma control questionnaire | 1month
  A simple questionnaire to measure the adequacy of asthma control and change in asthma control which occurs either spontaneously or as a result of treatment. 7 items; 1 week recall (for items on symptoms and rescue inhaler use). 7-point scale (0=no impairment, 6= maximum impairment for symptoms and rescue use; and 7 categories for FEV1%). Minimally important difference: Change in score of 0.5
Allergic rhinitis control test | Baseline
  It is 5-item questionnaire about the control of allergic rhinitis. Questions are scored from 1 to 5 and evaluated for rhinitis during the last 2 weeks. Total score between 5 and 25.
  ≥ 20: Good control of rhinitis; <20: Poor control of rhinitis
Allergic rhinitis control test | 1month
  It is 5-item questionnaire about the control of allergic rhinitis. Questions are scored from 1 to 5 and evaluated for rhinitis during the last 2 weeks. Total score between 5 and 25.
  ≥ 20: Good control of rhinitis; <20: Poor control of rhinitis
Fear of COVID-19 Scale | Baseline
  Bangla fear of COVID (FCV19-S): It is a questionnaire that assesses the fear of COVID-19. It consists of 7 items scored on a 5-item Likert scale. The higher the score, the more fear.
Fear of COVID-19 Scale | 1month
  Bangla fear of COVID (FCV19-S): It is a questionnaire that assesses the fear of COVID-19. It consists of 7 items scored on a 5-item Likert scale. The higher the score, the more fear.
COVID-19 Anxiety Scale (CAS) | Baseline
  Coronavirus anxiety scale (CAS): It is a scale that measures the anxiety generated by COVID-19 in the last two weeks. It presents 5 items and a score> 9 indicates dysfunctional anxiety associated with the pandemic.
COVID-19 Anxiety Scale (CAS) | 1month
  Coronavirus anxiety scale (CAS): It is a scale that measures the anxiety generated by COVID-19 in the last two weeks. It presents 5 items and a score> 9 indicates dysfunctional anxiety associated with the pandemic.
COVID Stress Scales | Baseline
  COVID stress scale (CSS): is a 36-item COVID Stress Scale (CSS) to measure these features, as they pertain to COVID-19. The CSS were developed to better understand and assess COVID-19-related distress. The scales were intentionally designed so they could be readily adapted for future pandemics.
COVID Stress Scales | 1month
  COVID stress scale (CSS): is a 36-item COVID Stress Scale (CSS) to measure these features, as they pertain to COVID-19. The CSS were developed to better understand and assess COVID-19-related distress. The scales were intentionally designed so they could be readily adapted for future pandemics.
Feeling of Satisfaction with Inhaler | Baseline
  This is a 10 items self-completed questionnaire to assess patient opinions regarding ease or difficulty of use, portability, and usability of devices for delivery of inhaled corticosteroids. The score ranges from 10-50 points. ≥ 43 points indicates high satisfaction; <43 points indicates low satisfaction
Feeling of Satisfaction with Inhaler | 1month
  This is a 10 items self-completed questionnaire to assess patient opinions regarding ease or difficulty of use, portability, and usability of devices for delivery of inhaled corticosteroids. The score ranges from 10-50 points. ≥ 43 points indicates high satisfaction; <43 points indicates low satisfaction
Test of Adherence to Inhalers | Baseline
  12-item questionnaire designed to assess the adherence to inhalers. The final version of the questionnaire included 12 items with two main domains, the patient (items #1 to #10) and the health professional (items #11 and #12) domain. In fact, the TAI consists of two complementary questionnaires: the 10-items TAI was designed to identify non-adherent patients and to establish the non-adherence level, whereas the 12-items TAI was designed to guide clinically the non-adherence patterns.An erratic and deliberate non-adherent behavioral pattern was defined in the presence of scores ≤24 for items #1 to #5 and items #6 to #10, respectively. The unwitting pattern was defined in the presence of a score 1 in at least one of the #11 or #12 items of the questionnaire.
Test of Adherence to Inhalers | 1month
  12-item questionnaire designed to assess the adherence to inhalers. The final version of the questionnaire included 12 items with two main domains, the patient (items #1 to #10) and the health professional (items #11 and #12) domain. In fact, the TAI consists of two complementary questionnaires: the 10-items TAI was designed to identify non-adherent patients and to establish the non-adherence level, whereas the 12-items TAI was designed to guide clinically the non-adherence patterns.An erratic and deliberate non-adherent behavioral pattern was defined in the presence of scores ≤24 for items #1 to #5 and items #6 to #10, respectively. The unwitting pattern was defined in the presence of a score 1 in at least one of the #11 or #12 items of the questionnaire.

IPD SHARING:
Plan to Share IPD: No